CLINICAL TRIAL: NCT04659707
Title: Evaluating Lung Structure and Function in Survivors of COVID-19 Using Hyperpolarized 129Xe MRI
Brief Title: Hyperpolarized 129Xe MRI of Survivors of COVID-19
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Peter J. Niedbalski, PhD, Research Assistant Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00146616
Record Dates: First submitted 2020-12-07; First posted 2020-12-09 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- COVID-19 Survivors (Experimental): Subjects recovering from COVID-19 disease will be imaged using hyperpolarized 129Xe MRI.
  Interventions: Drug: Hyperpolarized Xe129

INTERVENTIONS:
Drug: Hyperpolarized Xe129 — Subjects will inhale up to 4 doses of hyperpolarized Xenon gas in order to image pulmonary function.
  Other Names: HP Xenon; 129Xe

SUMMARY:
The purpose of this study is to evaluate pulmonary function of patients recovering from mild, moderate, and severe COVID-19 disease using hyperpolarized 129Xe MRI.

DETAILED DESCRIPTION:
COVID-19, the disease at the heart of the current global pandemic, is characterized by fevers, cough, sore throat, malaise, and myalgias, with 98% of patients experiencing some pulmonary involvement. In those infected with the causative virus, SARS-CoV-2, the severity of symptoms, as well as their duration, is widely variable. There is strong evidence from computed tomography (CT) images of patients with severe COVID-19 that pulmonary abnormalities and lung damage caused by infection may have long-term consequences for survivors. Furthermore, many patients with mild or moderate experience symptoms such as fatigue and dyspnea long (>60 days) after initial symptom onset, but there are currently no clinical predictors of which patients are at greatest risk for long-term health effects. As such, sensitive and specific predictors or biomarkers that can evaluate quality-of-life, risk of infection exacerbation, and long-term outcomes are critically needed.

Pulmonary imaging using hyperpolarized (HP) 129Xe magnetic resonance imaging (MRI) provides a means to detect abnormalities in the pulmonary small airways, vasculature, and parenchyma by quantifying pulmonary ventilation, gas diffusion, and regional gas exchange. HP 129Xe MRI is fast (<16s), non-invasive, and radiation free, making it a safe and effective method for characterizing lung function, even in individuals with lung disease. In this pilot study, we will use HP 129Xe to evaluate pulmonary structure and function in COVID-19 patients using the following specific aims:

Aim 1. Detect regional pulmonary function abnormalities in recovering COVID-19 patients using hyperpolarized 129Xe MRI. The hypothesis is that ventilation and gas exchange defects will be present in recovering COVID-19 patients, and further that the extent of impairment will correlate with disease severity.

Aim 2. Determine risk factors for long term outcomes using hyperpolarized 129Xe MRI and clinical biomarkers. The hypothesis is that HP 129Xe MRI biomarkers will predict long-term lung function impairment brought on by COVID-19.

These aims will be tested by performing HP 129Xe MRI in patients recovering from mild, moderate, or severe COVID-19. By coming to a fuller understanding of the long-term impairment of pulmonary function, future treatment can be optimized to minimize severe disease and health care utilization.

ELIGIBILITY:
Inclusion Criteria:

* Oxygenation saturation of ≥88% at rest by study staff within 48 hours prior to study entry.
* The participant has a previous diagnosis of COVID-19 confirmed by COVID-19 PCR or antibody testing and is being seen for outpatient follow-up.
* Subject is at least 10 days post-symptom-onset and do not have a fever (<99.5°).
* Ability to read and understand English or Spanish

Exclusion Criteria:

* Subject is less than 18 years old
* MRI is contraindicated based on responses to MRI screening questionnaire
* Subject is pregnant or lactating
* Subject does not fit into 129Xe vest coil used for MRI
* Subject cannot hold his/her breath for 15-16 seconds
* Subject deemed unlikely to be able to comply with instructions during imaging
* Oxygen saturation <88% on room air or with supplemental oxygen
* Cognitive deficits that preclude ability to provide consent
* Institutionalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Ventilation Defect Percentage | Baseline
  VDP at Baseline
Ventilation Defect Percentage | 6-months
  VDP at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified imaging data will be shared with researchers upon reasonable request.